CLINICAL TRIAL: NCT06927193
Title: Regional Analgesia at the Pediatric Emergency Department
Status: Not yet recruiting | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Neonatologist, Hillel Yaffe Medical Center
Other Study IDs: 0035-25-HYMC
Record Dates: First submitted 2025-04-06; First posted 2025-04-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Regional Anaesthesia
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Regional anaesthesia: Children who underwent regional analgesia during routine pediatric emergency department
  Interventions: Procedure: Regional anaesthesia

INTERVENTIONS:
Procedure: Regional anaesthesia — Regional anaesthesia

SUMMARY:
Approximately two years ago, ultrasound-guided regional blocks technique was introduced into routine use in the pediatric emergency department at Hillel Yaffe Medical Center. Since then, nearly 300 different blocks have been performed.

Study Objective: To collect a registry database of complication rates associated with regional analgesia during routine pediatric emergency department care between 2023 and 2025.

DETAILED DESCRIPTION:
Adequate pain management is a key component of pediatric emergency care. The use of regional analgesia, particularly ultrasound-guided regional blocks, has gained momentum in recent years as part of pain management, reducing the need for opioids and serving as a safe and effective alternative to procedural sedation.

For anesthesiologists, this is now a routine tool mainly performed in the operating room. In adult emergency medicine, this tool has also been integrated and is sometimes performed by emergency physicians.

In children, performing ultrasound-guided regional blocks presents additional challenges compared to adults. The primary challenge in an unsedated child is maintaining cooperation throughout the procedure. Other difficulties include limited maneuverability due to their smaller size, reduced allowable volume of local anesthetics (based on weight), and more. For these reasons, most ultrasound-guided regional blocks in children are performed in the operationg room after sedation or general anesthesia. There are only a few case reports describing the use of simple ultrasound-guided regional blocks performed by emergency physicians in pediatric ED settings.

Approximately two years ago, this technique was introduced into routine use in the pediatric emergency department at Hillel Yaffe Medical Center. Since then, nearly 300 different blocks have been performed.

Study Objective: To collect a registry database of complication rates associated with regional analgesia during routine pediatric emergency department care between 2023 and 2025.

ELIGIBILITY:
Inclusion Criteria:

* Children who visited the pediatric emergency department between 2023-2025 and underwent a nerve block during their visit.

Exclusion Criteria:

* Children who visited the emergency department but had the nerve block performed outside the emargency department setting (e.g., inpatient wards or operationg room), or if the block was performed by a physician not affiliated with the pediatric emergency department.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who visited the pediatric emergency department between 2023-2025
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Any complication | 2 years
  Any complication that happend to the patient because of the regional anaesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katzir Y, Ganor L, Berant R, Shahar-Nissan K. Building Blocks-A Block-by-Block Approach to Better Emergency Care in Children. Pediatr Emerg Care. 2024 Jun 1;40(6):463-468. doi: 10.1097/PEC.0000000000003201. Epub 2024 Apr 2. PMID 38563828
- [Background] Shahar-Nissan K, Berant R, Ganor L, Katzir Y. Ultrasound-Guided Supraclavicular Brachial Plexus Blocks Performed by Pediatric Emergency Medicine Physicians for Painful Orthopedic Procedures in a Pediatric Emergency Department-A Case Series. Pediatr Emerg Care. 2022 Dec 1;38(12):e1684-e1687. doi: 10.1097/PEC.0000000000002878. Epub 2022 Nov 18. PMID 36449743
- [Background] Ruest S, Anderson A. Management of acute pediatric pain in the emergency department. Curr Opin Pediatr. 2016 Jun;28(3):298-304. doi: 10.1097/MOP.0000000000000347. PMID 26974975
- [Background] Walker BJ, Long JB, Sathyamoorthy M, Birstler J, Wolf C, Bosenberg AT, Flack SH, Krane EJ, Sethna NF, Suresh S, Taenzer AH, Polaner DM, Martin L, Anderson C, Sunder R, Adams T, Martin L, Pankovich M, Sawardekar A, Birmingham P, Marcelino R, Ramarmurthi RJ, Szmuk P, Ungar GK, Lozano S, Boretsky K, Jain R, Matuszczak M, Petersen TR, Dillow J, Power R, Nguyen K, Lee BH, Chan L, Pineda J, Hutchins J, Mendoza K, Spisak K, Shah A, DelPizzo K, Dong N, Yalamanchili V, Venable C, Williams CA, Chaudahari R, Ohkawa S, Usljebrka H, Bhalla T, Vanzillotta PP, Apiliogullari S, Franklin AD, Ando A, Pestieau SR, Wright C, Rosenbloom J, Anderson T; Pediatric Regional Anesthesia Network Investigators. Complications in Pediatric Regional Anesthesia: An Analysis of More than 100,000 Blocks from the Pediatric Regional Anesthesia Network. Anesthesiology. 2018 Oct;129(4):721-732. doi: 10.1097/ALN.0000000000002372. PMID 30074928
- [Background] Frenkel O, Liebmann O, Fischer JW. Ultrasound-guided forearm nerve blocks in kids: a novel method for pain control in the treatment of hand-injured pediatric patients in the emergency department. Pediatr Emerg Care. 2015 Apr;31(4):255-9. doi: 10.1097/PEC.0000000000000398. PMID 25803747
- [Background] Baker MD, Gullett JP. Ultrasound-Guided Femoral Nerve Blocks. Pediatr Emerg Care. 2015 Dec;31(12):864-8; quiz 869-71. doi: 10.1097/PEC.0000000000000634. PMID 26626896
- [Background] Heffler MA, Brant JA, Singh A, Toney AG, Harel-Sterling M, Grandjean-Blanchet C, Riera A, Khalil PA, Starr-Seal RL, Binder ZW. Ultrasound-Guided Regional Anesthesia of the Femoral Nerve in the Pediatric Emergency Department. Pediatr Emerg Care. 2023 Feb 1;39(2):e30-e34. doi: 10.1097/PEC.0000000000002607. Epub 2022 Jan 12. PMID 35245015
- [Background] Argiris A, Heald P, Kuzel T, Foss FM, DiStasio S, Cooper DL, Arbuck S, Murren JR. Phase II trial of 9-aminocamptothecin as a 72-h infusion in cutaneous T-cell lymphoma. Invest New Drugs. 2001;19(4):321-6. doi: 10.1023/a:1010613912335. PMID 11561692